CLINICAL TRIAL: NCT06007105
Title: SUCCEED Africa: Protocol for a Multi-method Pilot Study of a Community-based Intervention for People With Psychosis in West and Southeast Africa
Brief Title: SUCCEED Africa: Support, Comprehensive Care and Empowerment of People With Psychosocial Disabilities
Acronym: SUCCEED
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: University of Ibadan (Other); University of Malawi (Other); University of Makeni (Unknown); University of Zimbabwe (Other); Zimbabwe National Association for Mental Health (ZIMNAMH) (Unknown); Mental Health Users and Carers Association (MeHUCA) Malawi (Unknown); The Asido Foundation (Unknown); Mental Health Coalition Sierra Leone (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 28346; EPPHZT74 (Other Grant/Funding Number: FCDO)
Record Dates: First submitted 2023-07-20; First posted 2023-08-23 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-07

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Schizotypal Disorder; Acute and Transient Psychotic Disorder; Delusional Disorder; Other Specified or Unspecified Primary Psychotic Disorder; Bipolar Type I Disorder With Psychotic Symptoms; Bipolar Type II Disorder With Psychotic Symptoms; Single Episode Depressive Disorder With Psychotic Symptoms; Recurrent Depressive Disorder With Psychotic Symptoms; Perinatal Mental or Behavioural Disorder With Psychotic Symptoms
Keywords: Sub-Saharan Africa; Psychosis; Co-Production; Peer support; Human rights; Nigeria; Malawi; Zimbabwe; Sierra Leone; Pilot trial; Schizophrenia; Community-based rehabilitation; Livelihoods
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Schizotypal Personality Disorder; Schizophrenia, Paranoid

STUDY DESIGN:
Intervention Model Description: This is a four-country pilot using a before-and-after study design to measure change in quality of life using the 26-item WHOQOL-BREF in participants with lived experience of psychosis who are offered the SUCCEED intervention (including case management, peer support and livelihoods activities) over a four-month follow-up period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SUCCEED Community-Based Intervention (Experimental): The SUCCEED community-based intervention (offering a combination of peer support, case management and livelihoods activities) will be delivered to 10 participants with lived experience of psychosis at each of the 4 pilot sites.
  Interventions: Behavioral: SUCCEED Community-Based Intervention

INTERVENTIONS:
Behavioral: SUCCEED Community-Based Intervention — The main components of the intervention are peer support, case management and livelihoods activities, delivered by a peer support worker and a community support worker. The peer support worker has lived experience of psychosis and draws on a variety of manualised tools and techniques adapted from previous studies. The community support worker mobilises families and communities to activate resources in support of participants (e.g., education and employment, social and recreational activities), drawing on established models of mental health case management and community-based inclusive development. The peer support worker and community support worker also run self-help groups for people with lived experience and their family members, respectively. Self-help group meetings are also used as an opportunity for group livelihoods activities taking an "ABCD" (asset-based community development" approach.

SUMMARY:
Although psychotic disorders typically affect less than 1% of the population, they are a significant cause of disability worldwide. Psychotic symptoms such as hallucinations, delusions and suicidal ideation can be profoundly disturbing, and negatively impact daily living. However, the social consequences of psychosis are often even more troubling than the symptoms. For example, people with psychosis have a high risk of experiencing violence, poverty, homelessness, incarceration, and unemployment, among other adverse outcomes.

There is a need for a range of accessible, appropriate interventions for people with psychosis to be delivered to those in the most vulnerable situations, including in low-resource settings in sub-Saharan Africa. A systematic review recently carried out as part of the formative research for SUCCEED identified 10 studies evaluating the impact of interventions for people with psychosis in Africa, most of which had a strongly clinical focus. The review concluded that there was a need for further research involving people with lived experience of psychosis in designing and evaluating holistic interventions that meet their diverse needs, within and beyond the health sector.

SUCCEED Africa is a six-year Health Research Programme Consortium (RPC) that has brought together people with lived experience of psychosis and people with professional experience (researchers, clinicians) from four African countries (Malawi, Nigeria, Sierra Leone, Zimbabwe) to co-produce a community-based intervention for psychosis, using a Theory of Change-driven approach. The SUCCEED intervention takes the World Health Organisation's (WHO's) CBR Matrix as a point of departure to consider the multifaceted needs of people living with psychosis and other psychosocial disabilities, and how best to meet these needs by mobilising the resources of individuals and families affected, as well as their broader communities.

This protocol describes a pilot study in which the SUCCEED intervention will be delivered and evaluated on a small scale, in preparation for a larger multi-country research evaluation using more rigorous methods, including randomised controlled trials in Nigeria and Zimbabwe and observational studies in Malawi and Sierra Leone, respectively. The main outcome of interest is change in subjective quality of life among participants with lived experience of psychosis who are offered the intervention over a four-month follow up period.

DETAILED DESCRIPTION:
Recognising the need for a framework for interventions to support people with psychosocial disabilities in LMICs, the WHO's 2010 CBR Guidelines included a special supplement on mental health, which drew mainly from expert opinion, evidence in community mental health, and basic development principles, to make recommendations for best practice. However, a 2016 review examining CBR for disabilities in LMICs identified only one example of CBR for psychosocial disabilities in Sub-Saharan Africa. The authors concluded that there was a need for more evidence from this region, in particular.

As part of SUCCEED Africa's formative research, a systematic review of the grey literature on CBR for psychosocial disabilities in LMICs was undertaken, in case there was in fact evidence available that had been excluded as a result of the previous review's strict eligibility criteria. The grey literature review identified 33 different CBR programmes, 11 of which were based in sub-Saharan Africa, but the quality of the evidence was generally very poor and too heterogeneous for any sort of meta-analysis. In contrast to previous reviews, the grey literature review found that the majority of programmes were not focused primarily on health, covering more domains of the CBR Matrix (e.g. livelihoods, empowerment, education, etc.). This suggests a disconnect between how CBR programmes are designed and evaluated to optimise clinical outcomes for research purposes, versus how they are designed to meet pragmatic needs in real-world practice.

The SUCCEED pilot will use a before-and-after study design looking at changes in subjective quality of life (WHOQOL-BREF) among participants with lived experience of psychosis who are offered the SUCCEED intervention over a four-month follow-up period. Key components of the SUCCEED intervention are peer support, case management and livelihoods activities, which are delivered by a gender-mixed team including one peer support worker and one community support worker embedded in a local organisation for persons with disabilities (OPD) in each SUCCEED country.

Nested within this pilot are three other components, described further in the full research protocol (available upon request) :

* A baseline assessment of the feasibility and acceptability of WHOQOL-BREF as a measurement tool (time taken to administer, proportion of participants who complete the tool, perspectives of data collectors assessed through interviews), face validity (assessed through cognitive interviewing) of WHOQOL-BREF, and the validity of proxy (completed by a close family member) versus self-completion.
* A qualitative study using a combination of focus groups (participants with psychosis, family members) and interviews (peer support workers, community support workers, supervisors, data collectors) to further examine the acceptability and feasibility of the SUCCEED's research and M&E tools (including WHOQOL-BREF) and processes.
* A process evaluation drawing on semi-structured observations and routine monitoring and evaluation (M&E) of intervention delivery, competency assessment of the two frontline providers (peer support workers and community support workers, via ENACT) research administrative data (adverse events, drop-outs), and end-line qualitative data (see above) to assess key process indicators and implementation outcomes (e.g. acceptability, appropriateness, feasibility, fidelity, safety, etc.).

ELIGIBILITY:
Inclusion criteria:

Participants with lived experience of psychosis must:

* Be consenting/assenting adults (age 18+)
* Be able to speak one of the main study languages: English, Chichewa, Krio, Shona, Yoruba
* Live within the pilot study area
* Have a current or past diagnosis of schizophrenia or other primary psychotic disorder, bipolar or depressive disorder with psychotic symptoms, or a maternal mental health or behavioural disorder with psychotic symptoms, as per the World Health Organisation's International Classification of Diseases Version 11 (see full list of eligible diagnoses, below).

For participants recruited from within the health care system, diagnosis will be confirmed from health records. For those identified in the community, a research worker will administer the World Health Organisation's Composite International Diagnostic Interview (WHO CIDI) screening tool for psychosis.

The following diagnoses are eligible for inclusion:

* Schizophrenia (6A20)
* Schizoaffective disorder (6A21)
* Schizotypal disorder (6A22)
* Acute and transient psychotic disorder (6A23)
* Delusional disorder (6A24)
* Other specified (6A2Y) or unspecified (6A2Z) primary psychotic disorder
* Bipolar type I disorder with psychotic symptoms (6A60.1, 6A60.5, 6A60.7, 6A60.A)
* Bipolar type II disorder with psychotic symptoms (6A61.3, 6A61.5)
* Single episode depressive disorder with psychotic symptoms (6A70.2, 6A70.4)
* Recurrent depressive disorder with psychotic symptoms (6A71.2, 6A71.4)
* Mental or behavioural disorder associated with pregnancy, childbirth or the puerperium, with psychotic symptoms (6E21)

Exclusion Criteria:

* People who are currently homeless, for logistical reasons; the SUCCEED intervention relies on PSWs and CSWs being able to regularly contact participants, including for home visits.
* People with secondary psychotic syndromes (6E61), as these are considered to be the direct consequences of physical health conditions as opposed to mental health conditions.
* People diagnosed with a substance-induced psychotic disorder (6C40.6-6C47.6), as recovery from substance use conditions is a specialist area outside the scope of the SUCCEED intervention under development.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-07-18 (Actual); Primary Completion 2023-12-15 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in self-reported Quality of Life (World Health Organisation Quality of Life Questionnaire Brief Version) | Baseline and at 4 months follow up (endpoint)
  WHOQOL-BREF has 26 items assessing individual's perception of their well-being over previous 2 weeks, across four domains (physical, psychological, social relationships and environment). Response to each item is rated against a 5-point Likert scale (1=not at all and 5=large amount). Scores are linearly transformed to total out of 100 where higher scores indicate better quality of life.
  WHOQOL-BREF may be administered by a data collector in an interview format or self-completed (with data collector available for any assistance needed). We will also invite a close family member to complete the WHOQOL-BREF independently at baseline to investigate reliability of self- versus proxy-reported quality of life. Both participants with lived experience of psychosis and family members will be asked to complete a cognitive interview checking understanding of the questionnaire following completion of the WHOQOL-BREF at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Professor Thomas Shakespeare, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (4):
- Kamuzu University of Health Sciences, Blantyre, Southern Region, Malawi
- University of Ibadan, Ibadan, Oyo State, Nigeria
- University of Makeni, Makeni, Northen Province, Sierra Leone
- University of Zimbabwe, Harare, North East, Zimbabwe

IPD SHARING:
Plan to Share IPD: Yes
Only anonymised data will be uploaded for archiving and data sharing. SUCCEED Data Access and Publication Policy stipulates that data are jointly owned by all SUCCEED partners; thus all partners are free to access anonymised SUCCEED data. Access is facilitated by the Data Management Team, which is comprised of nominated researchers at each site.
Supporting Information: Study Protocol
Time Frame: After an 18-month embargo period, data are prepared for upload to LSHTM Data Compass site, in line with FCDO UK guidance on data sharing.
Access Criteria: Any individual internal or external to SUCCEED may submit an expression of interest using a standardised online form outlining their intention to access and/or publish SUCCEED data; expressions of interest are reviewed on a regular basis by SUCCEED's five-country leadership team for approval. This is the main avenue by which SUCCEED ensures the use of data is for valid research. Once approved, those accessing the project data are required to sign a data access/confidentiality form.
URL: https://datacompass.lshtm.ac.uk/information.html

REFERENCES:
- [Background] Hunt X, Abdurahman H, Omobowale O, Afolayan A, Munetsi E, Dzapasi L, Mokaya N, Koroma A, Barrie I, Ogunmola O, Koroma A, Shakespeare T, Eaton J, Ryan G. Interventions for adolescents and adults with psychosis in Africa: a systematic review and narrative synthesis. Glob Ment Health (Camb). 2022 May 27;9:223-240. doi: 10.1017/gmh.2022.25. eCollection 2022. PMID 36618745
- [Background] Omigbodun OO, Ryan GK, Fasoranti B, Chibanda D, Esliker R, Sefasi A, Kakuma R, Shakespeare T, Eaton J. Reprioritising global mental health: psychoses in sub-Saharan Africa. Int J Ment Health Syst. 2023 Mar 28;17(1):6. doi: 10.1186/s13033-023-00574-x. PMID 36978186
- [Background] Bella-Awusah T, Abdurahman H, Omobowale O, Aturu O, Afolayan A, Ogunmola O, Fasoranti B, Olusanmi M, Tamambang R, Bamidele O, Ryan G, Shakespeare T, Eaton J, Omigbodun O. Lessons of Hope and Resilience: A Co-Produced Qualitative Study of the Experiences of Youth Living with Psychosis During the COVID-19 Pandemic in Nigeria. Community Ment Health J. 2024 Jan;60(1):47-59. doi: 10.1007/s10597-023-01128-8. Epub 2023 Jun 12. PMID 37306804
- [Background] Lee YY, Buyanga M, Mehta A, Omowunmi OA, Ryan G, Sunkel C, Vasquez A, Jones N. Cracks that Let the Light in: Collective Reflections on Integrating Lived Experience of Psychosis in Research and Policy in the Context of a Global Commission. Community Ment Health J. 2023 Jul;59(5):819-825. doi: 10.1007/s10597-023-01118-w. Epub 2023 Mar 20. PMID 36939989
- See also: Study webpage — https://www.lshtm.ac.uk/research/centres-projects-groups/succeed